CLINICAL TRIAL: NCT07321613
Title: Effect of Thalidomide, Carmofur and Compound Mylabris Capsules (TCC) Cocktail Combined With Transarterial Chemoembolization Versus Transarterial Chemoembolization Alone on Survival in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Effect of TCC Cocktail Combined With TACE Versus TACE Alone on Survival in uHCC Patients
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20251111101713560
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Cancer (HCC)
MeSH Terms: conditions — Liver Neoplasms | interventions — Thalidomide; carmofur

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TACE+cocktail: Patients in the TACE+cocktail group received TACE and took the combined oral medications daily, which consisted of thalidomide tablets, carmofur tablets , and compound mylabris capsule.
  Interventions: Drug: Thalidomide (50mg); Drug: carmofur; Drug: compound mylabris capsule; Procedure: TACE
- TACE only: Patients in the TACE only group received only TACE treatment.
  Interventions: Procedure: TACE

INTERVENTIONS:
Drug: Thalidomide (50mg) — Thalidomide tablets (Changzhou Pharmaceutical Factory, 50 mg qn)
  Groups: TACE+cocktail
Drug: carmofur — carmofur tablets (Qilu Pharmaceutical, 100 mg, tid)
  Groups: TACE+cocktail
Drug: compound mylabris capsule — CMC (Guizhou Yibai Pharmaceutical Co., Ltd, 750 mg, bid)
  Groups: TACE+cocktail
Procedure: TACE — received initial treatment with traditional TACE by well-trained and experienced physicians

SUMMARY:
This is a multicenter, retrospective cohort study that aims to evaluate the efficacy and safety of a triple-drug cocktail (TCC), consisting of Thalidomide, Carmofur, and Compound Mylabris Capsules (CMC), in combination with conventional Transarterial Chemoembolization (TACE) for the treatment of patients with unresectable Hepatocellular Carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* patients who met the HCC diagnostic criteria according to the Guidelines for Diagnosis and Treatment of Primary Liver Cancer in China.
* patients underwent conventional TACE.
* availability of complete medical records for data extraction and follow-up.

Exclusion Criteria:

* a history of previous or synchronous treatment for tumors such as radio frequency ablation (RFA) or systemic chemotherapy.
* poor liver functions (Child-Pugh class C).
* accompanying other life-threatening diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This multicenter, retrospective cohort study included adult patients (≥18 years old) diagnosed with unresectable hepatocellular carcinoma (HCC). The diagnosis was made according to the Chinese guidelines for the diagnosis and treatment of primary liver cancer (relevant edition). All patients received initial treatment with conventional transarterial chemoembolization (TACE).
Sampling Method: Non-Probability Sample
Enrollment: 545 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | up to five years
  Defined as the time interval from the date of the patient's first TACE treatment to the date of death from any cause or the date of the last follow-up (whichever occurred first).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) at 6 Months | up to six months
  The proportion of patients achieving a Complete Response (CR) or Partial Response (PR) according to mRECIST criteria at the 6-month follow-up after treatment initiation.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No